CLINICAL TRIAL: NCT01834716
Title: Exercise in Asymptomatic Pre-Alzheimer's Disease Pilot Study/ 18F-AV-45-A14 - CLINICAL EVALUATION OF FLORBETAPIR F 18 (18F-AV-45) Sponsor of 18F-AV-45-A14: Avid Radiopharmaceuticals
Brief Title: Exercise in Asymptomatic Pre-Alzheimer's Disease Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Neill R. Graff-Radford, M.D., M.D., Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 12-002817
Record Dates: First submitted 2013-04-15; First posted 2013-04-18 (Estimated); Results first posted 2019-03-29 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2018-12

CONDITIONS: Alzheimer's Disease Prevention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aerobics exercise (Experimental): Participants in this group will be randomized to aerobics exercise (the equivalent of walking briskly for 50 minutes three times per week).
  Interventions: Behavioral: Aerobic vs. Non-Aerobic exercise
- Non-Aerobics Exercise (Experimental): Participants in this group will be randomized to a non-aerobics (attending classes of toning and stretching a minimum of three times per week) exercise group.
  Interventions: Behavioral: Aerobic vs. Non-Aerobic exercise

INTERVENTIONS:
Behavioral: Aerobic vs. Non-Aerobic exercise

SUMMARY:
Researchers are trying to determine if cognitively normal subjects undergoing a moderate aerobic exercise program will accumulate less amyloid-ß (Aβ) concentration in their brain than subjects undergoing a non-aerobic exercise program, and further evaluating the safety and imaging characteristics of florbetapir F 18, the radioactive drug that will allow us to image changes in the brain amyloid-ß (Aβ).

DETAILED DESCRIPTION:
After screening assessments have been completed, subjects will be randomized into one of two groups: aerobic exercise group and non-aerobic exercise group. All subjects will be trained on the Physical Activity Scale for the Elderly (PASE), using the Body Media armband, and exercise diary. Subjects will also complete an online food questionnaire.

Subjects assigned to the aerobic exercise group will work with an exercise trainer who will provide individual training (six half hour sessions) until they are proficient at the use of the equipment and understand goals. Subjects will return to Brooks Family YMCA at their convenience, but at a minimum of four times per week. Subjects will complete the exercise journal daily and the Physical Activity Scale for the Elderly (PASE) questionnaire on a monthly basis.

Subjects assigned to the non-aerobic exercise group will attend supervised classes on toning and stretching at a minimum of four times per week. Subjects will complete the exercise journal daily and the Physical Activity Scale for the Elderly (PASE) questionnaire on a monthly basis.

ELIGIBILITY:
* 65 years of age or older.
* Not diagnosed with memory problems.
* Do not exercise in which you sweat and/or raise your pulse rate more than 30 minutes two times per week.
* Able to walk ten blocks (about one mile).
* Willing to participate in weekly exercise classes at the Brooks YMCA for six months.
* Able to have an MRI and CT/PET scan.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neill Graff-Radford, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited via study invitations mailed to persons by age and zip code. Local community presentations were also conducted to recruit subjects.
Groups:
- Non-Aerobics Exercise: Participants in this group will be randomized to a non-aerobics(attending classes of toning and stretching a minimum of three times per week) exercise group.
- Aerobics Exercise: Participants in this group will be randomized to an aerobics exercise group (the equivalent of walking briskly for 50 minutes three times per week).
Period: Overall Study
Arm/Group | Non-Aerobics Exercise | Aerobics Exercise
Started | 4 | 12
Completed | 4 | 11
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Non-aerobics Exercise: Participants in this group will be randomized to a non-aerobics exercise group (attending classes of toning and stretching a minimum of three times per week).
- Total: Total of all reporting groups
Arm/Group | Non-aerobics Exercise | Aerobics Exercise | Total
Number analyzed (Participants) | 4 | 12 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 4 | 12 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 1 | 8 | 9
Region of Enrollment [Number; unit: participants]
  United States | 4 | 12 | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Retained at 6 Months
Description: The number of subjects retained at 6 month end of study time point.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Aerobics Exercise: Participants in this group will be randomized to aerobics exercise.
  Aerobic vs. Non-Aerobic exercise
  12 enrolled 11 completed
- Non-Aerobics Exercise: Participants in this group will be randomized to a non-aerobics exercise group.
  Aerobic vs. Non-Aerobic exercise
  4 enrolled and 4 completed
Arm/Group | Aerobics Exercise | Non-Aerobics Exercise
Number analyzed (Participants) | 11 | 4
Participants | 11 | 4

ADVERSE EVENTS:
Time Frame: Adverse events were collected at baseline, 3 months, and 6 months.
Arm/Group | Aerobics Exercise | Non-Aerobics Exercise
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/12 | 0/4
Other Adverse Events (participants affected / at risk) | 0/12 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aerobics Exercise (N=12) | Non-Aerobics Exercise (N=4)
Cancer (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes